CLINICAL TRIAL: NCT01048905
Title: Phase 2 Trial for Glutamine Therapy for Hemolysis-Associated Pulmonary Hypertension
Brief Title: Glutamine Therapy for Hemolysis-Associated Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01FD003531-01 (FDA); IRB 2008-059 (Other: Institutional Review Board); 1R01FD003531-01 (FDA)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Hypertension; Sickle Cell Disease; Thalassemia
Keywords: Pulmonary Hypertension; Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell; Thalassemia | interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment: L-glutamine (Experimental): Patients will receive an 8-week course of oral L-glutamine 10 grams TID
  Interventions: Drug: L-Glutamine

INTERVENTIONS:
Drug: L-Glutamine — Oral L-glutamine 10 grams TID or (0.1g/kg TID) for children < 15 years of age.

SUMMARY:
The primary hypothesis of this study is that glutamine supplementation will improve the erythrocyte glutamine/glutamate ratio, a biomarker of oxidative stress, hemolysis and pulmonary hypertension (PH) in sickle cell disease (SCD) and thalassemia (Thal) patients with PH. PH is defined as a tricuspid regurgitant jet velocity (TRV) on Doppler echocardiography > 2.5 m/s. We also predict that glutamine therapy will increase arginine bioavailability and subsequently alter sickle red cell endothelial interaction that can be identified using endo-PAT technology through nitric oxide (NO) generation, leading to changes in biological markers, and clinical outcome. Specifically our second hypothesis is that oral glutamine will decrease biomarkers of hemolysis and adhesion molecules, and improve the imbalanced arginine-to-ornithine ratio that occurs in hemolytic anemias, leading to improved arginine bioavailability and clinical endpoints of endothelial dysfunction and PH in patients with SCD and Thal.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of SCD (Hb SS, SC or SBeta- thalassemia) or Thal
* PH documented by echocardiography, defined as at TRV greater than 2.5 m/s
* Age greater than or equal to 4 years

Exclusion Criteria:

* Inability to take or tolerate oral medication
* Acute crisis or hospitalization within 1 month of enrollment
* Hepatic dysfunction (SGPT greater than 3X normal)
* Renal dysfunction (Creatinine greater than 2X normal)
* Allergy to glutamine
* Pregnancy or breastfeeding
* Patients on sildenafil (Viagra), calcium channel blockers, or amino acid/protein supplements (other therapies acceptable if stable more than 3 months)

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Morris, MD, Principal Investigator — Emory University; Augusta Saulys, MD, Principal Investigator — Children's Hosptial & Research Center Oakland
Locations (1):
- Children's Hospital & Research Center Oakland, Oakland, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment: L-glutamine
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: L-glutamine
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Erythrocyte Glutamine/Glutamate Ratio [Mean (Standard Deviation); unit: Ratio] — Population: Blood work only available for N=6 participants, as reported here.
  Ratio
    number analyzed (Participants) | 6
    (all) | 1.75 (0.6)
Plasma Glutamine [Mean (Standard Deviation); unit: µmol/L] — Population: Blood work only available for N=6 participants, as reported here.
  µmol/L
    number analyzed (Participants) | 6
    (all) | 704.5 (137)
Tricuspid Regurgitant Jet Velocity on Doppler Echocardiography [Mean (Standard Deviation); unit: Meters per second] — Tricuspid Regurgitant Jet Velocity was measured using Doppler Echocardiography in meters per second.
  Meters per second | 3.0 (0.6)
6 Minute Walk Distance [Mean (Standard Deviation); unit: Meters] — The six-minute walk test (6MWT) measures the distance in meters an individual is able to walk over a total of six minutes on a hard, flat surface.
  Meters | 386 (94)
Liver Function Tests [Mean (Standard Deviation); unit: U/L]
  Alanine aminotransferase (ALT) | 40 (42)
  Aspartate aminotransferase (AST) | 73 (40)
Renal Function Tests [Mean (Standard Deviation); unit: mg/dL]
  Creatinine | 0.9 (0.4)
  Blood urea nitrogen (BUN) | 14 (10)

OUTCOME MEASURES:

1. Primary Outcome: Erythrocyte Glutamine/Glutamate Ratio at 8 Weeks
Description: Erythrocyte Glutamine/Glutamate Ratio: a novel biomarker of oxidative stress
Time Frame: 8 weeks
Population: Blood work only available for N=6 participants, as reported here.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment: L-glutamine
Number analyzed (Participants) | 6
Ratio | 2.40 (1.6)

2. Secondary Outcome: Plasma Glutamine
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Treatment: L-glutamine
Number analyzed (Participants) | 12
µmol/L | 685.8 (139)

3. Secondary Outcome: Tricuspid Regurgitant Jet Velocity on Doppler Echocardiography
Description: Tricuspid Regurgitant Jet Velocity was measured using Doppler Echocardiography in meters per second.
Time Frame: 8 week
Population: Data available for 11 participants only because one patient missed their appointment for their week 8 echocardiogram and was lost to follow up, and another patient died of sepsis before week 8 visit.
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Treatment: L-glutamine
Number analyzed (Participants) | 11
Meters per second | 2.8 (0.5)

4. Secondary Outcome: 6 Minute Walk Distance
Description: The six-minute walk test (6MWT) measures the distance in meters an individual is able to walk over a total of six minutes on a hard, flat surface.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Treatment: L-glutamine
Number analyzed (Participants) | 12
Meters | 366 (109)

5. Secondary Outcome: Liver Function Tests
Description: Alanine aminotransferase (ALT) Aspartate aminotransferase (AST)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment: L-glutamine
Number analyzed (Participants) | 12
U/L
  ALT | 38 (27)
  AST | 63 (26)

6. Secondary Outcome: Renal Function Tests
Description: Creatinine Blood urea nitrogen (BUN)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment: L-glutamine
Number analyzed (Participants) | 12
mg/dL
  Creatinine | 0.9 (0.3)
  BUN | 17 (7)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Treatment: L-glutamine
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: L-glutamine (N=13)
Pain (General disorders) | 3
Acute Chest Syndrome (General disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: L-glutamine (N=13)
Sexually Transmitted Disease Related Pain (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes